CLINICAL TRIAL: NCT03733977
Title: The Reliability And Validity Of Family Satisfaction In Intensive Care Unit 24 (FS-ICU 24) Scale In Turkish Language And The Evaluation Of ICU Patients' Relatives Satisfaction :An Observational Study
Brief Title: The Reliability And Validity Of Family Satisfaction In Intensive Care Unit 24 (FS-ICU 24) Scale In Turkish Language
Status: Completed | Type: Observational
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, ZEYNEP YUKSEL, Principal Investigator, TC Erciyes University
Other Study IDs: 2014/121
Record Dates: First submitted 2018-10-12; First posted 2018-11-07 (Actual); Last update posted 2018-11-07 (Actual); Status verified 2018-10

CONDITIONS: Family Satisfaction
Keywords: Family; Intensive Care Unit; Quality Of Care; Satisfaction
MeSH Terms: conditions — Personal Satisfaction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Purpose of this study was to investigate the validity and reliability of Family Satisfaction in the Intensive Care Unit-24 (FC-ICU 24) survey in Turkish language, evaluation the satisfaction of intensive care unit patients' relatives and to determine the factors affecting satisfaction.

DETAILED DESCRIPTION:
Family Satisfaction in the Intensive Care Unit-24 (FC-ICU 24) survey is valid and reliable survey which was used to evaluate family satisfaction of intensive care units.

Turkish version which was prepared based on FS-ICU 24 survey was applied to the relatives of ICU patients (the ICUs in Anesthesiology, Internal Medicine, General Surgery and Neurosurgery ) in the Erciyes University Medical Faculty. The study was conducted between April and June 2015. The Turkish version was tested for reliability and validity, and it was proven to be reliable and valid. The subjects of the study were relatives of patients that were hospitalized for at least 48 hours, who had visited the patient at least once. Only one relative was included in the study per patient, and the survey was conducted after the required permissions were taken from the related medical departments.

ELIGIBILITY:
Inclusion Criteria:

* Family member of intensive care unit patient ( at least 48 hours hospitalization) aged at least 18

Exclusion Criteria:

* Rejection of family member

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Family members of intensive care unit patients at least 48 hours hospitalization.
Sampling Method: Non-Probability Sample
Enrollment: 369 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Family Satisfaction in Intensive Care Unit (FS-ICU 24) Survey Validation In Turkish Language | An Average Of 3 Months
  Family Satisfaction in Intensive Care Unit (FS-ICU 24) Survey was shown to demonstrate family satisfaction from intensive care units effectively. The survey evaluated the following topics: treatment, care, the attitudes of the ICU staff, environmental conditions, the decision-making process. We evaluate the reliability and the validity of the FS-ICU 24 survey in the Turkish language for demonstrate cross cultural adaptation of survey. The Turkish version ( that was prepared based on the FS-ICU 24 survey ) applied to the relatives of patients who were hospitalized for at least two days and had visited the patient at least once in tertiary intensive care units. The answers to the survey questions ranged from excellent (1 point) to poor (5 points), consistent with the original survey. The results ranged from 20 to 100 points. 20 points indicated excellent satisfaction, 100 points indicated poor satisfaction. The satisfaction decreases as the score increases.

CONTACTS AND LOCATIONS:
Overall Officials: ZEYNEP YUKSEL TURHAN, M.D., Principal Investigator — Sanliurfa Education and Research Hospital; AYNUR AKIN, PROF., Study Director — ERCIYES UNIVERSITY MEDICAL FACULTY
Locations (1):
- Sanliurfa Education and Research Hospital, Sanliurfa, Turkey (Türkiye)